CLINICAL TRIAL: NCT06224595
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetic, Pharmacodynamic Profiles Following Single and Multiple Doses and Food Effect of CS32582 Capsules in Healthy Adult Subjects
Brief Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetic, Pharmacodynamic Profiles and Food Effect of CS32582 Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS32582-101
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-01

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: The study consists of 3 parts: single ascending dose (SAD), food effect (FE) and multiple ascending dose (MAD). Both SAD and MAD study are a randomized, double-blind, placebo-controlled dose-escalation design. The FE study is a randomized, open-label, two-period, two-crossover design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- CS32582 Cohort 1 (Experimental): Subjects receive a single dose of 3 mg CS32582 or matching placebo
  Interventions: Drug: CS32582 capsule; Drug: Placebo capsule
- CS32582 Cohort 2 (Experimental): Subjects receive a single dose of 6 mg CS32582 or matching placebo
  Interventions: Drug: CS32582 capsule; Drug: Placebo capsule
- CS32582 Cohort 3 (Experimental): Subjects receive a single dose of 12 mg CS32582 or matching placebo
  Interventions: Drug: CS32582 capsule; Drug: Placebo capsule
- CS32582 Cohort 4 (Experimental): Subjects receive a single dose of 24 mg CS32582 or matching placebo
  Interventions: Drug: CS32582 capsule; Drug: Placebo capsule
- CS32582 Cohort 5 (Experimental): Subjects receive a single dose of 36 mg CS32582 or matching placebo
  Interventions: Drug: CS32582 capsule; Drug: Placebo capsule
- CS32582 Cohort 6 (Experimental): Subjects receive a single dose of 54 mg CS32582 or matching placebo
  Interventions: Drug: CS32582 capsule; Drug: Placebo capsule
- CS32582 Cohort 7 (Experimental): Subjects receive a single dose 12 mg CS32582 in either the fasted or fed state for two periods
  Interventions: Drug: CS32582 capsule
- CS32582 Cohort 8 (Experimental): Subjects receive 3 mg CS32582 or matching placebo for 10 days, twice daily (every 12 h) from Day 1 to Day 9, and once on Day 10.
  Interventions: Drug: CS32582 capsule; Drug: Placebo capsule
- CS32582 Cohort 9 (Experimental): Subjects receive 6 mg CS32582 or matching placebo for 10 days, twice daily (every 12 h) from Day 1 to Day 9, and once on Day 10.
  Interventions: Drug: CS32582 capsule; Drug: Placebo capsule
- CS32582 Cohort 10 (Experimental): Subjects receive 12 mg CS32582 or matching placebo for 10 days, once daily from Day 1 to Day 10.
  Interventions: Drug: CS32582 capsule; Drug: Placebo capsule
- CS32582 Cohort 11 (Experimental): Subjects receive 12 mg CS32582 or matching placebo for 10 days, twice daily (every 12 h) from Day 1 to Day 9, and once on Day 10.
  Interventions: Drug: CS32582 capsule; Drug: Placebo capsule

INTERVENTIONS:
Drug: CS32582 capsule — Participants receive CS32582 orally single or multiple doses
Drug: Placebo capsule — Participants receive placebo matching CS32582 orally single or multiple doses
  Arms: CS32582 Cohort 1; CS32582 Cohort 10; CS32582 Cohort 11; CS32582 Cohort 2; CS32582 Cohort 3; CS32582 Cohort 4; CS32582 Cohort 5; CS32582 Cohort 6; CS32582 Cohort 8; CS32582 Cohort 9

SUMMARY:
The study is to evaluate the safety, tolerability, pharmacokinetic and pharmacodynamic profiles of CS32582 after single or multiple oral administration, as well as the food effect on the pharmacokinetics in healthy subjects.

DETAILED DESCRIPTION:
This study consists of 3 parts: single ascending dose (SAD), food effect (FE) and multiple ascending dose (MAD). Both SAD and MAD study are randomized, double-blind, placebo-controlled design. The FE study is a randomized, open-label, two-period, two-crossover design.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects, both male and female.
* Between18 and 55 years of age (inclusive) at screening visit.
* BMI between 19.0-26.0 kg/m^2 (including critical value) at screening visit and baseline visit, male subjects' body weight ≥ 50 kg, female subjects' body weight ≥45 kg.
* Subject is medically healthy or judged by the investigator to be abnormal but clinically insignificant based on the results of history inquiry, physical examination, vital signs, standard 12-lead electrocardiogram, X-ray, abdominal ultrasound examination, and clinical laboratory tests at the time of screening visit.
* All subjects and female partners of male agree to use medically recognized effective methods of contraception (including physical contraception, surgical contraception, abstinence, etc.) from the start of signing informed consent form to 3 months after the last dose.
* Subjects voluntarily participate in the study and sign informed consent form.

Exclusion Criteria:

* History of clinically significant drug allergy or atopic allergic diseases (asthma, urticaria, eczematous dermatitis) or drug allergy to investigational products or similar investigational products.
* History of cardiovascular system, endocrine system, nervous system, respiratory system, digestive system, liver, kidney, blood and lymphatic system, immune system, psychiatric diseases and metabolic abnormalities.
* Conditions that may affect the determination of skin adverse events related to the investigational drug, including but not limited to sunburn, excessive tattooing (covering more than 25% of body surface area), or existing acne extending beyond sebum-prone areas (i.e., arms, torso, back, buttocks, and/or genital area).
* History of myalgia or rhabdomyolysis.
* History of hereditary hyperbilirubinemia.
* History of gastrointestinal, hepatic, or renal diseases or surgeries within the past 6 months that could affect drug absorption or metabolism, excluding uncomplicated appendectomy and hernia repair.
* History of active tuberculosis or positive tuberculosis at the screening visit.
* History of recurrent bacterial, fungal, or viral infections (≥3 occurrences in the past year, excluding common cold), or active infection requiring treatment at the screening visit, or history of infection within ≤8 weeks before baseline visit requiring intravenous anti-infective drugs and/or hospitalization, or history of infection requiring oral anti-infective drugs ≤2 weeks before baseline visit.
* Untreated diarrhea at baseline visit or diarrhea symptoms within 7 days before the planned first dose.
* History of drug abuse.
* Vaccination within the past 3 months at the screening visit or plans for any vaccination during the study.
* Participation in an interventional clinical trial (device or drug) within the past 3 months or use of investigational drugs within the past 3 months or still within 5 half-life of that drug (whichever is longer) at the screening visit.
* Blood donation or significant blood loss (>300 mL) within the past 3 months at the screening visit.
* Use of any prescription drugs, non-prescription drugs, any vitamin products, or herbal products within the past month before baseline visit.
* Inability to tolerate venepuncture or history of needle or blood-related fainting.
* Regular alcohol consumption exceeding 7 drinks per week for females or 14 drinks per week for males in the past 3 months at the screening visit, or use of any alcohol-containing product within 48 hours before the planned first dose.
* Smoking more than 5 cigarettes or equivalent tobacco daily within the past 3 months at the screening visit or inability to quit smoking during the study.
* Consumption of excessive tea, coffee, and/or caffeine-containing beverages (more than 8 cups) daily within the past 14 days before baseline visit, or consumption of tea, coffee, and/or caffeine-containing beverages or foods within 48 hours before the planned first dose.
* Consumption of grapefruit or grapefruit-containing products within the past 14 days before baseline visit.
* Systolic blood pressure less than 90 mmHg or greater than 140 mmHg, and/or diastolic blood pressure less than 60 mmHg or greater than 90 mmHg at screening and baseline visits.
* Glomerular filtration rate (eGFR) <90 mL/min (calculated using CKD-EPI equation with blood creatinine, age, and gender) at screening and baseline visits.
* QTcF ≥450 ms or other clinically significant abnormalities of standard 12-lead electrocardiogram judged by the investigator at screening and baseline visits.
* Meeting any of the following at screening and baseline visits: Blood routine: White blood cell count <3.5×10^9/L or neutrophil count <1.8×10^9/L or hemoglobin <115 g/L for females or <130 g/L for males; or platelet count <125×10^9/L. Blood creatinine above the upper limit of normal (ULN). Alanine aminotransferase or aspartate aminotransferase or total bilirubin or direct bilirubin above ULN.
* Inability to provide a negative human immunodeficiency virus (HIV) antibody report at screening visit.
* Positive results for syphilis serology, hepatitis B surface antigen (HBsAg), HBV-DNA quantification, or hepatitis C virus antibody (HCV-Ab) at screening and baseline visits.
* Positive urine drug abuse screening (opiates, methamphetamine, ketamine, ecstasy, marijuana, cocaine) or positive alcohol breath test at screening and baseline visits.
* Pregnant or lactating females, or females with serum human chorionic gonadotropin (HCG) ≥5 mIU/mL.
* Need or plan to engage in strenuous physical activity or exercise during the study.
* Participants unable to tolerate a high-fat meal (applicable only to participants in postprandial trials).
* Participants with swallowing difficulties.
* Other situations deemed unsuitable for participation in the clinical trial by the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Incidence and Severity of Adverse Events (AEs) | From the time of signing the informed consent form to 7 days after the last administration of the drug
  To investigate the safety and tolerability by assessment of AEs following administration.
Pharmacokinetic parameters - Area Under the Curve(AUC) | From time 0 to 48 hours for single dose. From time 0 to 48 hours after the last dose for multiple doses. From time 0 to 48 hours after each period's dosing for food effect study.
  Area Under the Plasma Concentration-time Curve of CS32582.
Pharmacokinetic parameters - Peak Plasma Concentration (Cmax) | From time 0 to 48 hours for single dose. From time 0 to 48 hours after the last dose for multiple doses. From time 0 to 48 hours after each period's dosing for food effect study.
  Maximum Observed Plasma Concentration of CS32582.
Pharmacokinetic parameters - Time of Peak Concentration(Tmax) | From time 0 to 48 hours for single dose. From time 0 to 48 hours after the last dose for multiple doses. From time 0 to 48 hours after each period's dosing for food effect study.
  Time to reach maximum observed plasma concentration of CS32582.
Pharmacokinetic parameters - Plasma Elimination Half-Life(t1/2) | From time 0 to 48 hours for single dose. From time 0 to 48 hours after the last dose for multiple doses. From time 0 to 48 hours after each period's dosing for food effect study.
  Plasma Elimination Half-Life of CS32582.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No